CLINICAL TRIAL: NCT02645656
Title: Topical Application of Curcumin Incorporated in Orabase in OSMF Patients
Brief Title: Topical Application of Curcumin Orabase in Oral Submucous Fibrosis (OSMF)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: SVS Institute of Dental Sciences (Other)
Responsible Party: Principal Investigator, Dr R Viswa Chandra, Ethics Committee Investigator, SVS Institute of Dental Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SVSIDS/OMR/EX1/2013
Record Dates: First submitted 2015-12-29; First posted 2016-01-05 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Oral Submucous Fibrosis
Keywords: Oral Submucous Fibrosis; Curcumin
MeSH Terms: conditions — Oral Submucous Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Curcumin Arm (Experimental): Curcumin gel will be applied in sites with Oral Submucous Fibrosis at designated time intervals.
  Interventions: Drug: Curcumin Arm

INTERVENTIONS:
Drug: Curcumin Arm — Curcumin gel will be applied in sites with Oral Submucous Fibrosis at designated time intervals

SUMMARY:
Curcumin (diferuloylmethane) is the chief component of the spice turmeric and is derived from the rhizome of the East Indian plant Curcuma longa. Curcuma longais a member of the Zingiberacae (ginger) family of botanicals and is a perennial plant that is native to Southeast Asia. Turmeric contains a class of compounds known as the curcuminoids, comprised of curcumin, demethoxy curcumin and bisdemethoxycurcumin.

DETAILED DESCRIPTION:
Anti-inflammatory mechanisms implicated in the anticarcinogenic potential of curcumin include: (1) inhibition of NF-κB and COX-2 (increased levels of COX-2 are associated with many cancer types); (2)inhibition of arachidonic acid metabolism via lipoxygenase and scavenging of free radicals generated in this pathway; (3) decreased expression of inflammatory cytokines IL-1b, IL-6, and TNF-a, resulting in growth inhibition of cancer cell lines; and (4) down-regulation of enzymes, such as protein kinase C, that mediate inflammation and tumor-cell proliferation.

Curcumin's potent anti-oxidant and free-radical quenching properties play an important role in the inhibitory effects of the compound on the initial stages of carcinogenesis. Antioxidants are implicated in the pathogenesis of OSMF and hence this preparation may be helpful in resolution of this lesion.

ELIGIBILITY:
Inclusion Criteria:

* Subjects showing classic clinical signs of OSMF and not under any intervention for the same will be included.

Exclusion Criteria:

* Subjects who are receiving or have received any form of therapy in the six month period leading to the study will be excluded.

Ages: 22 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-12; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Reduction in OSMF lesion | up to 6 months
  The number of bands and the consistency of the lesion will be evaluated at designated time intervals using appropriate indices.

SECONDARY OUTCOMES:
Jaw Opening | up to 6 months
  Jaw opening in mm will be measured at designated time intervals using an appropriate instrument.

CONTACTS AND LOCATIONS:
Overall Officials: Ramaraju Devaraju, MDS, Study Director — Academic Commitee
Locations (1):
- SVS Institute of Dental Sciences, Mahabubnagar, Hyderabad, Andhra Pradesh, India

IPD SHARING:
Plan to Share IPD: No
Data will be released after publishing the findings.